CLINICAL TRIAL: NCT02107456
Title: The Long Term Effect of Dry Needling on Myofascial Trigger Point in the Upper Trapezius Muscle.
Brief Title: Effect of Dry Needling on Myofascial Trigger Point
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Social Welfare and Rehabilitation Science (Other)
Responsible Party: Principal Investigator, Amir Massoud Arab, Dr., University of Social Welfare and Rehabilitation Science
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: 920114
Record Dates: First submitted 2014-04-03; First posted 2014-04-08 (Estimated); Last update posted 2014-04-08 (Estimated); Status verified 2014-04

CONDITIONS: Pain
Keywords: Dry Needling, Myofascial trigger point, Upper trapezius
MeSH Terms: conditions — Pain | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dry Needling (Experimental): The taut band of trigger point in upper trapezius muscle; localized between the thumb and index finger, was needled forward and backward repeatedly until there were no more local twitch response
  Interventions: Device: Dry Needling

INTERVENTIONS:
Device: Dry Needling — Dry needling was performed for one week, three times a week.
  Other Names: Western Accupuncture

SUMMARY:
Myofascial trigger point is one of the most common causes of musculoskeletal disorders. Myofascial trigger point in upper trapezius has been reported as a symptom in patients with neck and upper thoracic pain. The purpose of this study was to investigate the prolonged effect of dry needling on myofascial trigger point in upper trapezius muscle.

DETAILED DESCRIPTION:
Pain intensity and Disability of arm, hand and shoulder (DASH) were collected at base line and at the end of treatment sessions, two weeks and three months follow up in both groups.

ELIGIBILITY:
Inclusion Criteria:

* 1. Presence of a palpable taut band in muscle.
* 2. Presence of a hypersensitive tender spot in the taut band.
* 3. Reproduction of the typical referred pain pattern of the MTP in response to compression. To detect active TrPs, TrP pressure tolerance was assessed using a mechanical pressure algometer. The investigator applied continuous pressure with the algometer with an approximate pressure of 2.5 kg/cm2.
* 4. Spontaneous presence of the typical referred pain pattern and/or patient recognition of the referred pain as familiar.
* 5- Pain of at least 30 mm on a visual analogue scale (VAS). The selected MTP of the UT muscle was located in the middle of the more nearly horizontal fibers of the UT 40.

Exclusion Criteria:

* had a history of fibromyalgia syndrome, whiplash injury, cervical spine surgery and fracture, cervical radiculopathy, having therapy within the past month before the study
* any systematic disease such as rheumatism and tuberculosis or cervical myelopathy, multiple sclerosis
* local infection,
* pregnancy
* taking anticoagulants (e.g. warfarin)
* long-term steroid using

Ages: 20 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 33 (Actual)
Dates: Start 2012-07; Primary Completion 2013-02 (Actual); Study Completion 2013-06 (Actual)

PRIMARY OUTCOMES:
Pain intensity | One year
  Pain intensity using visual analogue scale (VAS) were collected at base line and at the end of treatment.

SECONDARY OUTCOMES:
Disability | One year
  Disability of Arm and Shoulder was collected at base line and at the end of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Amir M Arab, PhD, Principal Investigator — University of Social Welfare and Rehabilitation Sciences
Locations (1):
- University of Social Welfare and Rehabilitation Sciences, Tehran, Tehran Province, Iran